CLINICAL TRIAL: NCT04613843
Title: Cold Water Immersion Stirring in Hyperthermic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Riana Pryor, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003720
Record Dates: First submitted 2020-10-30; First posted 2020-11-03 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Hyperthermia
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Intervention Model Description: Randomized, counterbalanced, crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water stirring (Active Comparator)
  Interventions: Other: Water Stirring
- No water stirring (Experimental)
  Interventions: Other: No Water Stirring

INTERVENTIONS:
Other: Water Stirring — Following an active heating protocol, the cooling intervention includes vigorous water stirring throughout cold water immersion.
  Arms: Water stirring
Other: No Water Stirring — Following an active heating protocol, the cooling intervention includes no water stirring throughout cold water immersion.
  Arms: No water stirring

SUMMARY:
The best way to cool a very hot person is using cold water immersion, however, the optimization of this technique has not been established. The goal of this study is to determine differences in cooling rates among two types of cold water immersion and passive cooling following immersion.

ELIGIBILITY:
Inclusion Criteria:

* 18-39 y old men and women
* Self-reported to be healthy
* Currently completes aerobic exercise at least 30 minutes a day, at least 2 days per week

Exclusion Criteria:

* History of any cardiovascular, neurologic, renal, or metabolic disease
* History of any contraindications on the CoreTemp contraindications and warnings document
* Current tobacco use or regular use within the last 2 years
* Taking medications with known thermoregulatory or cardiovascular effects (e.g., aspirin, beta blockers, diuretics, psychotropics, etc.)
* History of exertional heat stroke
* Currently pregnant or breastfeeding
* Inability to follow the rules of the protocols or understand the consent form

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Cooling rate | 20 minutes
  The core temperature cooling rate

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Research and Exercise in Special Environments, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be made available upon written request.